CLINICAL TRIAL: NCT02018835
Title: Exercise Stress MRI to Evaluate Aortic Function (Compliance, Distensibility, Pulse Wave Velocity) and Left Ventricular Function : Validation in Healthy Volunteers and in Selected Patients. A Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012-A01093-40; 2012-28 (Other: AP HM)
Record Dates: First submitted 2012-11-26; First posted 2013-12-23 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- patients of an insufficiency organic severe surgical mitrale (Other)
  Interventions: Device: MRI; Device: cardiac echography transthoracic
- insufficiency organic mitrale moderated in severe asymptomatic (Other)
  Interventions: Device: MRI; Device: cardiac echography transthoracic
- patients of an aortic bicuspidie (Other)
  Interventions: Device: MRI; Device: cardiac echography transthoracic
- patients of a syndrome of Marfan (Other)
  Interventions: Device: MRI; Device: cardiac echography transthoracic
- Healthy volunteers (Other)
  Interventions: Device: MRI; Device: cardiac echography transthoracic

INTERVENTIONS:
Device: MRI
Device: cardiac echography transthoracic

SUMMARY:
Detecting abnormalities in the left ventricular mechanical and hemodynamic response to the stress of exercise may offer early diagnostic indicators in patients suffering from valvular disease such as mitral regurgitation. Ultrasound-based imaging methods have been gaining importance in providing prognosis among those patients. However, decreased signal to noise ratio in the images and increased motion-related artifacts during exercise stress echocardiography have been reported, with a lack of reproducibility of results and a the limitation of its availability only in reference centers. In our laboratory, we are able to perform supine bicycle exercise MRI (1.5 T) using the Lode ergometer mounted on the far end of the patient table, previously described in healthy volunteers.

The first aim of our study is to demonstrate the safety and the feasibility of our MRI protocol in selected patients with asymptomatic severe organic mitral regurgitation, to assess left ventricular volumes and function, and regurgitant volume in comparison to exercise cardiac echography.

Besides, few recent studies sustain the relevance of novel markers of central aortic function (compliance, distensibility and pulse wave velocity) assessed by noninvasive MRI to explore vascular aging. In monogenic connective tissue diseases, altered arterial stiffness is the premature signature of the disease in asymptomatic patients. Noninvasive evaluation of aortic stiffness would be useful for risk assessment and preventive follow-up strategies in young asymptomatic relatives of subjects with aortic inherited diseases, such as syndromic and non-syndromic familial forms of thoracic aortic aneurysm and /or dissection. Furthermore, this technique should be able to evaluate the effect of drugs on aortic stiffness change in trials, before and after drug therapy, more relevant than the classic change in aortic diameter measurement.

The second aim of our study is 1) to provide the sensibility of our MRI protocol to estimate local and regional heterogeneity in aortic functional parameters (distensibility, compliance and PWV) 2) to evaluate the predictive value of these regional aortic parameters assessed by MRI to diagnose and to stratify the aortopathy related to presymptomatic Marfan patients and to bicuspid aortic valve in young adults, in comparison to carotids-femoral pulse wave velocity estimation by applanation tonometry.

ELIGIBILITY:
Inclusion Criteria:

* Autonomous ADULT patient,

patient Marfan:

* under their usual treatment(processing) (including ß blocking)
* diagnosis confirmed by the molecular biology (transfer(transformation) of the gene FBN1)
* Asymptomatic or Dilation of the aorta = 40 mm on the ascending aorta on an echocardiography or an imaging in cups(cuttings) dating less than 6 months.

PATIENT Aortic bicuspid :

* Diagnosis confirmed by cardiac echography and/or imaging in cups(cuttings)
* Asymptomatic or Dilation of the aorta = 40 mm on the ascending aorta, and absence of valvulopathy aortic significant (IA of rank I in II, absence of significant RA), on the echocardiography or the imaging in cups(cuttings) dating less than 6 months.

patients Insufficiency mitral organic moderated in severe asymptomatic:

* SOR > 30 mm2, on an echocardiography or an imaging in cups(cuttings) dating less than 6 months
* Absence of ischemic or functional cause
* Patient recovering from a functional evaluation by echography of effort

patients Insufficiency mitral organic severe surgical

* SOR > 40 mm2, on an echocardiography or an imaging in cups(cuttings) dating less than 6 months
* Absence of ischemic or functional cause
* Status functional: stage(stadium) II of the NYHA
* Patient recovering from a functional evaluation by echography of effort

Volunteer healthy :

* affiliated to the Social Security
* having given its agreement by signed consent
* not presenting contraindication to the realization of a MRI

Exclusion Criteria:

* Patient claustrophobic,
* patient refusing the protocol or the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-12-05 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
blood samples | 24 MONTHS
  to estimate local and regional heterogeneity in aortic functional parameters

SECONDARY OUTCOMES:
aortic function | 24 MONTHS
  MRI - magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique Hopitaux De Marseille; alexis jacquier, Principal Investigator — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France